CLINICAL TRIAL: NCT06963853
Title: Evaluation of Microbial and Endocrinological Parameters in Dialysis Patients With Sepsis
Status: Recruiting | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Etty Kruzel-Davila, Head of the Nephrology Department, Western Galilee Hospital-Nahariya
Other Study IDs: 0086-22-NHR
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sepsis; Hemodialysis
Keywords: blood cultures; parathyroid hormone; catheter; infection; cardiovascular; mortality
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodialysis patients with suspected catheter-related bloodstream infections (CRBSIs).: Study Population:
  The study will include hemodialysis patients over the age of 18 who are hospitalized at the Galilee Medical Center due to sepsis and have provided written informed consent to participate in this study.
  Study Procedure:
  During hospitalization, and as part of the clinical workup for sepsis, blood cultures will be obtained from three sources:
  1. The central venous catheter (CVC),
  2. The dialysis machine circuit, and
  3. A peripheral vein. In addition, parathyroid hormone (PTH) levels will be measured through a blood sample.
  Interventions: Diagnostic Test: Blood cultures will be obtained from three sources: 1. The central venous catheter (CVC), 2. The dialysis machine circuit, and 3. A peripheral vein

INTERVENTIONS:
Diagnostic Test: Blood cultures will be obtained from three sources: 1. The central venous catheter (CVC), 2. The dialysis machine circuit, and 3. A peripheral vein — PTH levels during sepsis and compare them to baseline pre-infection levels, with serial follow-up of PTH values post-recovery.

SUMMARY:
This prospective study aims to evaluate the diagnostic value and reliability of blood cultures obtained from different sources-central venous catheter (CVC), dialysis machine, and peripheral vein-in hemodialysis patients with suspected catheter-related bloodstream infections (CRBSIs). By comparing the timing and rates of bacterial growth from each site, the study seeks to identify the most accurate and timely method for diagnosing bloodstream infections in this patient population.

In addition, the study will assess the dynamics of parathyroid hormone (PTH) levels during acute infections. Specifically, it will investigate whether a significant drop in PTH levels-and the rate of recovery following infection-correlates with adverse outcomes such as infectious complications, cardiovascular morbidity, or 90-day mortality. These findings may offer valuable prognostic insights and support improved monitoring and treatment strategies for dialysis patients experiencing infection.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a major global public health challenge, affecting millions of individuals worldwide. A significant proportion of these patients progress to end-stage kidney disease (ESKD), necessitating renal replacement therapies such as hemodialysis (HD). Beyond the gradual decline in renal function, CKD is associated with a high burden of comorbidities, particularly cardiovascular disease (CVD) and infections .Patients with CKD undergoing hemodialysis are especially vulnerable to infections, which represent a major contributor to morbidity and mortality in this population. This increased susceptibility is largely attributable to secondary immunodeficiency associated with kidney disease (SIDKD), the repeated need for vascular access, and the presence of multiple coexisting conditions.

Vascular access through catheters, grafts, or fistulas is essential for dialysis treatment. According to the 2023 USRDS report, in 2021, over 85% of individuals who began hemodialysis initiated treatment using a central venous catheter (CVC). Patients undergoing hemodialysis with a central venous catheter (CVC) are at increased risk for catheter-related bloodstream infections (CRBSIs), which are associated with significant morbidity, including a higher incidence of cardiovascular events, increased mortality, and substantial healthcare costs.6-10 The incidence of catheter-related infections has been reported to range from 1.1 to 5.5 episodes per 1,000 CVC days.

A retrospective study reported a median time of 163 days to the first episode of CRBSI.13 Several studies have identified a range of risk factors associated with CRBSI in hemodialysis patients. These include diabetes mellitus, age under 75 years, prolonged use of tunneled or implanted catheters, immunosuppressive therapy, colonization with methicillin-resistant Staphylococcus aureus (MRSA), and a history of bacteremia or bacteriuria within three months prior to catheter insertion. Additional factors include dialysis vintage, the site of catheter placement, number of catheterizations and abnormal laboratory parameters such as low albumin, elevated C-reactive protein (CRP), and reduced hemoglobin levels.

Diagnosis of CRBSI is challenging, as not all bacteremia in dialysis patients originates from catheters.

Diagnosis requires at least 1 positive blood culture from a peripheral source (dialysis circuit or vein) and no other apparent source, with either positive semiquantitative (>15 CFU/ catheter segment, hub or tip) or quantitative (>102 CFU/catheter segment, eg, hub or tip) culture, whereby the same organism (species and antibiogram) is isolated from the catheter segment (eg, hub or tip) and a peripheral source (dialysis circuit or vein) blood sample. If available, the following would be supportive: Simultaneous quantitative cultures of blood samples with a ratio of ≥3:1 (catheter hub/tip vs peripheral [dialysis circuit/vein]); differential period of catheter culture versus peripheral BC positivity of 2 hours. According to the Centers for Disease Control and Prevention (CDC), a compatible clinical presentation, along with at least one positive peripheral blood culture and no other identifiable source of infection, combined with growth of the same organism from a tunneled catheter tip, either positive semiquantitative culture (>15 CFU/catheter segment) or quantitative culture (>10³ CFU/catheter segment), supports the diagnosis of a catheter-related infection.

However, peripheral venous access is often limited in dialysis patients due to the need to preserve veins for future vascular access creation. Due to the challenges associated with obtaining peripheral venous blood samples, a study conducted in Canada compared the results of peripheral blood cultures to cultures taken from tunneled catheters and from the dialysis machine during treatment. This study demonstrated that blood cultures drawn from the dialysis circuit during treatment had higher sensitivity and specificity for detecting catheter-related bloodstream infections compared to peripheral blood cultures. Despite these findings, current guidelines for evaluating catheter-related bloodstream infections have not changed, and there is still a recommendation to obtain catheter hub/tip vs peripheral [dialysis circuit/vein]).

Parathyroid hormone (PTH) may influence immune function, yet data on PTH fluctuations during infections in dialysis patients are limited. Studies suggest low PTH levels are associated with recurrent infections and increased mortality.

Fluctuations in parathyroid hormone (PTH) levels during infection may be driven by elevated levels of pro-inflammatory cytokines such as IL-6 and IL-1β, which upregulate the expression of calcium-sensing receptors (CaSR) on the parathyroid gland, thereby leading to suppressed PTH secretion.

In critically ill patients, including those with septic shock or extensive burns, hypocalcemia has been frequently observed. This phenomenon may be partially explained by the presence of high extracellular calcium concentrations in necrotic tissues, which can stimulate pro-inflammatory cytokine release and activate the CaSR, contributing to inflammation-induced hypocalcemia. Notably, CaSR has been proposed to function as a chemokine-like receptor, promoting inflammatory responses and cytokine recruitment.

In addition to its role in calcium-phosphate homeostasis, PTH is known to modulate immune function. Elevated PTH levels promote T-lymphocyte proliferation and IL-2 secretion, whereas suppressed PTH levels-particularly below 65 pg/mL-have been associated with reduced CD4/CD8 ratios and increased susceptibility to infections in dialysis patients.

Moreover, low PTH levels have been linked to malnutrition and the development of malnutrition-inflammation complex syndrome (MICS), a condition commonly observed in the dialysis population.

Despite the biological rationale outlined above, it remains unclear whether PTH levels fluctuate during infection and whether such changes carry prognostic significance. A clinical observation in the dialysis unit at the Galilee Medical Center led to the hypothesis that PTH levels decrease during episodes of sepsis.

This study aims to characterize whether a significant decline in PTH levels occurs during sepsis, while simultaneously evaluating additional metabolic parameters such as white blood cell count, hemoglobin, platelets, calcium, phosphate, albumin, and CRP. Furthermore, we plan to assess the rate of PTH recovery following clinical resolution of infection and explore its potential association with clinical outcomes, including recurrent infections, cardiovascular morbidity, and mortality.

Research Hypothesis:

1. In hemodialysis patients with catheter-related bloodstream infections, blood cultures drawn from the dialysis machine are expected to detect infection as effectively, or possibly more effectively, than peripheral venous blood cultures.
2. Changes in parathyroid hormone (PTH) levels may indicate an increased risk of mortality, potentially informing treatment adjustments and monitoring strategies in dialysis patients with acute infections.

Study Objectives:

1. To compare the diagnostic yield of blood cultures obtained from three different sources in hemodialysis patients:

   * Central venous catheter (CVC),
   * Dialysis machine (during treatment),
   * Peripheral vein.
2. To measure PTH levels during sepsis and compare them to baseline pre-infection levels, with serial follow-up of PTH values post-recovery.
3. To assess clinical outcomes including infectious and cardiovascular complications, and mortality, in correlation with PTH levels in patients experiencing sepsis.

ELIGIBILITY:
Inclusion Criteria: hemodialysis patients over the age of 18 who are hospitalized at the Galilee Medical Center due to sepsis and have provided written informed consent to participate in this study.

-

Exclusion Criteria: • Patients with cognitive impairment who are unable to provide informed consent.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients over the age of 18 who are hospitalized at the Galilee Medical Center due to sepsis and have provided written informed consent to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Positive Blood Cultures by Sampling Site Among Documented Bloodstream Infections (CVC, Dialysis Machine, Peripheral Vein) | Within 21 days of hospitalization
  This outcome measure will compare the proportion of positive blood cultures obtained from three different sampling sites-central venous catheter (CVC), dialysis machine, and peripheral vein-among all confirmed cases of bloodstream infection in dialysis patients. The goal is to evaluate the diagnostic yield of each site and identify the most sensitive and reliable source for detecting bloodstream infections. Findings will support evidence-based recommendations regarding the preferred site for blood culture collection in this population. Comparative analysis will include statistical evaluation of sensitivity, yield, and agreement between sites.
Change in Parathyroid Hormone (PTH) Levels During Infection and Rate of PTH Recovery Post-Discharge | 90 days post-discharge
  This outcome measure will evaluate the change in parathyroid hormone (PTH) levels during acute infection and the monthly rate of recovery after hospital discharge in dialysis patients. PTH levels will be measured at three time points: (1) during the acute infection, (2) at discharge, and (3) monthly for up to 90 days post-discharge. The primary analysis will assess the magnitude of PTH suppression during infection and the trajectory of recovery over time. These parameters will be analyzed for their correlation with key 90-day outcomes, including infectious complications, cardiovascular events, and all-cause mortality. Statistical analyses will include repeated measures ANOVA and mixed-effects models to evaluate longitudinal changes and their association with clinical endpoints.

SECONDARY OUTCOMES:
Rate of Recurrent Infections Within 90 Days of Hospital Discharge | 90 days post-discharge
  This secondary outcome will assess the rate of recurrent infections occurring within 90 days of hospital discharge among dialysis patients who experienced an initial infectious episode. The analysis will examine whether the magnitude of PTH suppression during infection and the rate of PTH recovery post-discharge are associated with the risk of recurrent infection. Recurrent infections will be defined based on clinical and microbiological criteria. Statistical analysis will include logistic regression and time-to-event models.
Incidence of Cardiovascular Events Within 90 Days of Hospital Discharge | 90 days post-discharge
  This secondary outcome will assess the incidence of cardiovascular events occurring within 90 days of discharge among dialysis patients following an infectious episode. The analysis will explore whether the degree of parathyroid hormone (PTH) suppression during infection and the rate of PTH recovery are associated with cardiovascular risk. Cardiovascular events will include acute coronary syndrome, arrhythmia, stroke, and heart failure exacerbation, confirmed by clinical documentation. Statistical models such as Cox proportional hazards or logistic regression will be used to evaluate associations.
All-Cause Mortality Within 180 Days of Hospital Discharge. | 180 days post-discharge
  This secondary outcome will evaluate all-cause mortality within 180 days following hospital discharge in dialysis patients who experienced an infectious episode. The analysis will investigate whether the extent of parathyroid hormone (PTH) suppression during infection and the rate of PTH recovery post-discharge are associated with mortality risk. Deaths will be confirmed through clinical records or national registries. Cox proportional hazards models will be used to assess the relationship between PTH dynamics and mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Galilee Medical Center, Nahariya, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
The following individual participant data (IPD) will be shared:
  Demographic information (age, sex, dialysis vintage)
  Clinical data relevant to the study (reason for hospitalization, comorbidities, dialysis modality)
  Blood culture results from all sampling sites (central catheter, dialysis machine, peripheral vein)
  Laboratory values, including PTH levels at baseline and during infection
  Outcome data, including complications during hospitalization, cardiovascular events, and 90-day mortality
  All shared data will be de-identified to protect patient confidentiality, in compliance with relevant privacy regulations and ethical guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual participant data (IPD) and supporting information will be available beginning 6 months after publication of the primary results and will remain available for 5 years thereafter.
Access Criteria: The individual participant data (IPD) and supporting documentation will be available beginning six months after publication of the study results in a peer-reviewed journal.
  Data will remain available for a period of five years following that date. A direct link to the IPD access page will be provided on the Galilee Medical Center website upon publication of the study results."
URL: https://www.gmc.org.il

REFERENCES:
- [Background] Dukkipati R, Kovesdy CP, Colman S, Budoff MJ, Nissenson AR, Sprague SM, Kopple JD, Kalantar-Zadeh K. Association of relatively low serum parathyroid hormone with malnutrition-inflammation complex and survival in maintenance hemodialysis patients. J Ren Nutr. 2010 Jul;20(4):243-54. doi: 10.1053/j.jrn.2009.10.006. Epub 2010 Mar 3. PMID 20199875
- [Background] Ozdemir FN, Yakupoglu U, Turan M, Arat Z, Karakayali H, Erdal R, Turan M. Role of parathormone levels on T-cell response in hemodialysis patients. Transplant Proc. 2002 Sep;34(6):2044-5. doi: 10.1016/s0041-1345(02)02846-4. No abstract available. PMID 12270308
- [Background] Canaff L, Zhou X, Hendy GN. The proinflammatory cytokine, interleukin-6, up-regulates calcium-sensing receptor gene transcription via Stat1/3 and Sp1/3. J Biol Chem. 2008 May 16;283(20):13586-600. doi: 10.1074/jbc.M708087200. Epub 2008 Mar 17. PMID 18348986
- [Background] Hendy GN, Canaff L. Calcium-sensing receptor, proinflammatory cytokines and calcium homeostasis. Semin Cell Dev Biol. 2016 Jan;49:37-43. doi: 10.1016/j.semcdb.2015.11.006. Epub 2015 Nov 21. PMID 26612442
- [Background] Hong YA, Kim JH, Kim YK, Chang YK, Park CW, Kim SY, Kim YS, Kang SW, Kim NH, Kim YL, Yang CW. Low parathyroid hormone level predicts infection-related mortality in incident dialysis patients: a prospective cohort study. Korean J Intern Med. 2020 Jan;35(1):160-170. doi: 10.3904/kjim.2018.264. Epub 2019 Oct 28. PMID 31648433
- [Background] Quittnat Pelletier F, Joarder M, Poutanen SM, Lok CE. Evaluating Approaches for the Diagnosis of Hemodialysis Catheter-Related Bloodstream Infections. Clin J Am Soc Nephrol. 2016 May 6;11(5):847-854. doi: 10.2215/CJN.09110815. Epub 2016 Apr 1. PMID 27037271
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee (HICPAC) (Appendix 1). Summary of recommendations: Guidelines for the Prevention of Intravascular Catheter-related Infections. Clin Infect Dis. 2011 May;52(9):1087-99. doi: 10.1093/cid/cir138. No abstract available. PMID 21467014
- [Background] Guo H, Zhang L, He H, Wang L. Risk factors for catheter-associated bloodstream infection in hemodialysis patients: A meta-analysis. PLoS One. 2024 Mar 27;19(3):e0299715. doi: 10.1371/journal.pone.0299715. eCollection 2024. PMID 38536779
- [Background] Delistefani F, Wallbach M, Muller GA, Koziolek MJ, Grupp C. Risk factors for catheter-related infections in patients receiving permanent dialysis catheter. BMC Nephrol. 2019 May 31;20(1):199. doi: 10.1186/s12882-019-1392-0. PMID 31151433
- [Background] Hoen B, Paul-Dauphin A, Hestin D, Kessler M. EPIBACDIAL: a multicenter prospective study of risk factors for bacteremia in chronic hemodialysis patients. J Am Soc Nephrol. 1998 May;9(5):869-76. doi: 10.1681/ASN.V95869. PMID 9596085
- [Background] Murea M, James KM, Russell GB, Byrum GV 3rd, Yates JE, Tuttle NS, Bleyer AJ, Burkart JM, Freedman BI. Risk of catheter-related bloodstream infection in elderly patients on hemodialysis. Clin J Am Soc Nephrol. 2014 Apr;9(4):764-70. doi: 10.2215/CJN.07710713. Epub 2014 Mar 20. PMID 24651074
- [Background] Martin K, Lorenzo YSP, Leung PYM, Chung S, O'flaherty E, Barker N, Ierino F. Clinical Outcomes and Risk Factors for Tunneled Hemodialysis Catheter-Related Bloodstream Infections. Open Forum Infect Dis. 2020 Apr 11;7(6):ofaa117. doi: 10.1093/ofid/ofaa117. eCollection 2020 Jun. PMID 32550235
- [Background] Shingarev R, Barker-Finkel J, Allon M. Natural history of tunneled dialysis catheters placed for hemodialysis initiation. J Vasc Interv Radiol. 2013 Sep;24(9):1289-94. doi: 10.1016/j.jvir.2013.05.034. Epub 2013 Jul 18. PMID 23871694
- [Background] Lok CE, Foley R. Vascular access morbidity and mortality: trends of the last decade. Clin J Am Soc Nephrol. 2013 Jul;8(7):1213-9. doi: 10.2215/CJN.01690213. PMID 23824198
- [Background] Ravani P, Gillespie BW, Quinn RR, MacRae J, Manns B, Mendelssohn D, Tonelli M, Hemmelgarn B, James M, Pannu N, Robinson BM, Zhang X, Pisoni R. Temporal risk profile for infectious and noninfectious complications of hemodialysis access. J Am Soc Nephrol. 2013 Oct;24(10):1668-77. doi: 10.1681/ASN.2012121234. Epub 2013 Jul 11. PMID 23847278
- [Background] Foley RN, Guo H, Snyder JJ, Gilbertson DT, Collins AJ. Septicemia in the United States dialysis population, 1991 to 1999. J Am Soc Nephrol. 2004 Apr;15(4):1038-45. doi: 10.1097/01.asn.0000119144.95922.c4. PMID 15034107
- [Background] Foley RN. Infections and cardiovascular disease in patients with chronic kidney disease. Adv Chronic Kidney Dis. 2006 Jul;13(3):205-8. doi: 10.1053/j.ackd.2006.04.006. PMID 16815226
- [Background] Ravani P, Quinn R, Oliver M, Robinson B, Pisoni R, Pannu N, MacRae J, Manns B, Hemmelgarn B, James M, Tonelli M, Gillespie B. Examining the Association between Hemodialysis Access Type and Mortality: The Role of Access Complications. Clin J Am Soc Nephrol. 2017 Jun 7;12(6):955-964. doi: 10.2215/CJN.12181116. Epub 2017 May 18. PMID 28522650
- [Background] Lok CE, Huber TS, Lee T, Shenoy S, Yevzlin AS, Abreo K, Allon M, Asif A, Astor BC, Glickman MH, Graham J, Moist LM, Rajan DK, Roberts C, Vachharajani TJ, Valentini RP; National Kidney Foundation. KDOQI Clinical Practice Guideline for Vascular Access: 2019 Update. Am J Kidney Dis. 2020 Apr;75(4 Suppl 2):S1-S164. doi: 10.1053/j.ajkd.2019.12.001. Epub 2020 Mar 12. PMID 32778223
- [Background] Johansen KL, Gilbertson DT, Li S, Li S, Liu J, Roetker NS, Ku E, Schulman IH, Greer RC, Chan K, Abbott KC, Butler CR, O'Hare AM, Powe NR, Reddy YNV, Snyder J, St Peter W, Taylor JS, Weinhandl ED, Wetmore JB. US Renal Data System 2023 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2024 Apr;83(4 Suppl 1):A8-A13. doi: 10.1053/j.ajkd.2024.01.001. No abstract available. PMID 38519262
- [Background] Steiger S, Rossaint J, Zarbock A, Anders HJ. Secondary Immunodeficiency Related to Kidney Disease (SIDKD)-Definition, Unmet Need, and Mechanisms. J Am Soc Nephrol. 2022 Feb;33(2):259-278. doi: 10.1681/ASN.2021091257. Epub 2021 Dec 14. PMID 34907031
- [Background] Bello AK, Okpechi IG, Osman MA, Cho Y, Htay H, Jha V, Wainstein M, Johnson DW. Epidemiology of haemodialysis outcomes. Nat Rev Nephrol. 2022 Jun;18(6):378-395. doi: 10.1038/s41581-022-00542-7. Epub 2022 Feb 22. PMID 35194215
- [Background] Bello AK, Alrukhaimi M, Ashuntantang GE, Basnet S, Rotter RC, Douthat WG, Kazancioglu R, Kottgen A, Nangaku M, Powe NR, White SL, Wheeler DC, Moe O. Complications of chronic kidney disease: current state, knowledge gaps, and strategy for action. Kidney Int Suppl (2011). 2017 Oct;7(2):122-129. doi: 10.1016/j.kisu.2017.07.007. Epub 2017 Sep 20. PMID 30675426
- [Background] Francis A, Harhay MN, Ong ACM, Tummalapalli SL, Ortiz A, Fogo AB, Fliser D, Roy-Chaudhury P, Fontana M, Nangaku M, Wanner C, Malik C, Hradsky A, Adu D, Bavanandan S, Cusumano A, Sola L, Ulasi I, Jha V; American Society of Nephrology; European Renal Association; International Society of Nephrology. Chronic kidney disease and the global public health agenda: an international consensus. Nat Rev Nephrol. 2024 Jul;20(7):473-485. doi: 10.1038/s41581-024-00820-6. Epub 2024 Apr 3. PMID 38570631